CLINICAL TRIAL: NCT00826982
Title: Minimally Invasive Detection of Lymphatic Micrometastases in Pancreatic Cancer
Acronym: Sonoma
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 07-006640; MCR SPORE (CA102701-05DJ); ACG (FNDT-1)
Record Dates: First submitted 2009-01-20; First posted 2009-01-22 (Estimated); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pancreatic Cancer

SUMMARY:
The major goal of this project is to reduce unnecessary pancreatic resections, namely resection in those patients with non-regional lymph node metastatses that cannot be cured with surgical resection. By combined minimally invasive methods for non-surgical biopsy and highly sensitive molecular assays for cancer cells, we believe we can increase the ability to detect distant lymph node metastases prior to surgical resection, and direct those patients for more appropriate therapy (including possible neo-adjuvant chemotherapy with or without surgery). We hypothesize that the combination of EUS-FNA and polymerase chain reaction (PCR) of a multimarker panel will increase the sensitivity for malignant lymph nodes compared with EUS-FNA cytology in patients with pancreatic ductal adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a mass in the pancreas suspicious for adenocarcinoma without biopsy proven distant metastases.
* Patients who are scheduled for clinically indicated EUS

Exclusion Criteria:

* Patients who are medically unfit for endoscopic sedation or surgery due to severe comorbid disease such as uncontrolled coronary disease, or oxygen dependant pulmonary disease.
* Patients who have any other malignancy other than basal cell carcinoma within the past 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Care
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2008-01; Primary Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
To determine the if molecular biomarkers increase the sensitivity by at least 5% for detection of malignant lymph nodes in patients with pancreatic ductal adenocarcinoma as compared to EUS-FNA cytology of lymph nodes alone. | End of study

SECONDARY OUTCOMES:
To determine the degree of RNA overexpression of pancreas cancer specific biomarkers in the pre-operative fine needle aspirate of lymph nodes and tumors of patients with pancreatic cancer using a set of pancreas cancer specific biomarkers | End of study

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wallace, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Jacksonville, Florida, United States